CLINICAL TRIAL: NCT02116348
Title: Effect of Nerve Growth Factor (Cerebrolysin) Therapy on Neurodevelopment, Sleep Pattern and Quality of Life in Children With Traumatic Brain Injury and Cerebral Palsy
Brief Title: Cerebrolysin Neural Repair Therapy in Children With Traumatic Brain Injury and Cerebral Palsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWA 000017585
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Cerebral Palsy Children; Children With Traumatic Brain Injury; Mental Handicap; Delayed Speech Development
Keywords: Cerebral palsy children; Cerebrolysin; Sleep questionnaire; Quality of life; Bayley III scale
MeSH Terms: conditions — Language Development Disorders | interventions — cerebrolysin; Nerve Growth Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cerebrolysin (Experimental): Nerve growth factor Cerebrolysin will be given to the intervention group
  Interventions: Drug: Cerebrolysin (Nerve growth factor)
- Conventional (No Intervention): These children will receive conventional treatment for cerebral palsy

INTERVENTIONS:
Drug: Cerebrolysin (Nerve growth factor) — Cerebrolysin will be given to the intervention group
  Other Names: Cerebrolysin
  Arms: Cerebrolysin

SUMMARY:
Cerebral palsy (CP) is the most frequent cause of motor handicap among children. The economic burden of CP in USA includes $1.18 billion in direct medical costs, $1.05 billion in direct non-medical costs, and an additional $9.24 billion in indirect costs, for a total cost of $11.5 billion or $921,000 average cost per person. Associated disabilities as mental retardation, delayed speech development add psychological burden of the disease on the family as well as economic burden.

Mental retardation is the major problem in children with cerebral palsy. Improving mental development will have a positive effect on quality of life for the child and his family. Treating associated impairments (mental retardation) with Cerebrolysin will improve mental development and quality of life, and will decrease the economic burden in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy with mental retardation
* Severe perinatal brain insult

Exclusion Criteria:

1. Severe growth retardation
2. Gastrostomy tube feeding
3. Intractable seizures.
4. Severe motor handicap and deformities from long standing spasticity.
5. Congenital malformations.
6. Suspected inborn error of metabolism.
7. Suspected inherited neurologic disease.
8. Children with auditory and visual impairments.
9. Care giver's refusal to participate in the study.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
neurodevelopment | 6 months
  Intelligence quotient (IQ) assessment at base line and after 3 and 6 month of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M.A. Hassanein, MD, PhD, Principal Investigator — Pediatric Department, Children's Hospital, Faculty of Medicine, Ain Shams University
Locations (1):
- Pediatric Department, Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Abassia, Egypt

REFERENCES:
- See also: Faculty of Medicine, Ain Shams University — http://med.asu.edu.eg/
- See also: Ain Shams University web site — http://www.asu.edu.eg/